CLINICAL TRIAL: NCT06859645
Title: Effects of Telerehabilitation-Based Motor Imagery Training on Pain, Trunk Endurance, Functional Capacity, and Psychosocial Parameters in People With Non-Specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Motor Imagery Training in Non-Specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hilal Karakas, M.Sc., Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MotorImagery
Record Dates: First submitted 2025-02-21; First posted 2025-03-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: telerehabilitation; motor imagery; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor Imagery and Exercise Group (Experimental): Participants in the intervention group will follow a pre-designed motor imagery program in addition to the prescribed exercise training for eight weeks. This program will include exercise videos specifically targeting the lumbar region, along with synchronized audio recordings providing detailed explanations of the exercises. The exercise videos will initially consist of simple exercises and will progressively advance to more complex movements over the course of the intervention. Participants will receive new exercise videos weekly. Each session will last approximately 20-25 minutes, and participants will be required to complete the program daily.
  Interventions: Behavioral: Motor imagey training; Behavioral: Exercise training
- Exercise Group (Active Comparator): Participants in the control group will receive only telerehabilitation-based exercise training under the supervision of a physiotherapist, twice a week for eight weeks.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Motor imagey training — In addition to the prescribed exercise training, participants in the intervention group will follow a pre-designed motor imagery program for eight weeks, practicing daily. This program will include pre-recorded exercise videos specifically targeting the lumbar region, along with synchronized audio recordings providing detailed explanations of the exercises.
  Arms: Motor Imagery and Exercise Group
Behavioral: Exercise training — All participants will receive telerehabilitation-based exercise training under the supervision of a physiotherapist for eight weeks. The exercise program will be delivered via videoconferencing as part of a telerehabilitation-based approach. The exercises, conducted under the physiotherapist's supervision, will consist of flexibility and stabilization exercises targeting the lumbar region and will last approximately 25 minutes per session.

SUMMARY:
Low back pain is a significant global health issue, affecting a large proportion of the population at some point in their lives. Among the different types of low back pain, non-specific low back pain is the most common. Chronic low back pain has been shown to impact trunk endurance, functional capacity, fatigue, anxiety, and depression levels.

Neuroscience-based studies aimed at improving pain management have demonstrated that chronic pain is associated with not only peripheral changes but also central changes. These central changes include abnormalities in the distribution of sensory cortical processing, disinhibition of the motor cortex, and disturbances in body schema perception.

Studies have shown that motor imagery training, defined as the mental simulation of movement without actual execution, functions as a cortical-level training method and has positive effects on impaired body schema perception, thereby reducing pain. A review of the literature indicates that motor imagery training contributes to the treatment of pathological pain syndromes such as complex regional pain syndrome, brachial plexus avulsion injury, phantom limb pain, distal radius fracture, and stroke by modulating cortical mechanisms. However, no randomized controlled trials have investigated the effectiveness of adding motor imagery training to exercise therapy in individuals with non-specific chronic low back pain, specifically regarding its impact on physical function and psychosocial parameters.

The aim of this study is to investigate the effects of a motor imagery training protocol, applied in addition to exercise therapy, on pain, physical, and psychosocial parameters in individuals with non-specific chronic low back pain.

A total of 32 individuals with chronic non-specific low back pain will be included in the study. Participants will be randomly assigned to either the intervention or control group. All participants will receive telerehabilitation-based exercise therapy under the supervision of a physiotherapist. In addition to the exercise therapy, participants in the intervention group will undergo asynchronous motor imagery training every day for eight weeks, while the control group will receive only exercise therapy.

Assessments will be conducted three times: before treatment, at the end of the 8-week intervention, and at the 12th week follow-up. All assessments will be performed through a telerehabilitation-based approach. The study will evaluate participants' pain, fatigue, disability level due to low back pain, anxiety and depression levels, and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 55 years old
* Having a history of low back pain persisting for at least three months
* Experiencing recurrent episodes of low back pain
* Having a low back pain intensity score of 4 or higher on the Numeric Pain Rating Scale (NRS) out of 10 during both rest and activity
* Having the ability to use a computer, tablet, or smartphone at a level sufficient to participate in assessments and treatment sessions via videoconference, or having a caregiver who can assist with this
* Volunteering to participate in the study
* Being able to read and understand Turkish

Exclusion Criteria:

* A history of spinal surgery
* Having traumatic low back injuries
* Presence of severe comorbidities (neurological, neuromuscular, cardiological, psychiatric)
* Presence of tumoral conditions
* Having visual or hearing impairments
* Presence of cognitive impairments
* Receiving physiotherapy for low back pain within the last six months
* Changes in pain medication within the last two months
* Receiving additional treatments beyond routine care
* Being pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Scale | Baseline, at 8 week, at 12 week
  The severity of general low back pain experienced by the participants in the last two days will be assessed numerically using the Numeric Pain Scale. Participants will be informed that a score of 0 represents "no pain at all," while a score of 10 represents "the most unbearable pain." Pain severity will be recorded numerically on a scale from 0 to 10.

SECONDARY OUTCOMES:
Oswestry Disability Index | Baseline, at 8 week, at 12 week
  The "Oswestry Disability Index" will be used to assess the level of disability related to low back pain among participants. This index evaluates the impact of low back pain on daily activities through 10 questions, each scored between 0 and 5, covering aspects such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and changes in pain severity. A lower score indicates a higher quality of life. The validity and reliability of the Turkish version of the index have been established, with a reported Cronbach's alpha of 0.91.
Fatigue Severity Scale | Baseline, at 8 week, at 12 week
  The "Fatigue Severity Scale," commonly used in clinical and experimental studies, will be employed to determine participants' fatigue levels. The scale consists of nine questions, each scored from 1 to 7 (1: strongly disagree, 7: strongly agree). The total score is obtained by summing the scores of all items and calculating the average. Higher scores indicate greater fatigue. This scale was developed and adapted into Turkish.
Hospital Anxiety and Depression Scale | Baseline, at 8 week, at 12 week
  The "Hospital Anxiety and Depression Scale" will be used to evaluate participants' levels of anxiety and depression. This scale is utilized to determine the risk, severity, and level of anxiety and depression in individuals. The HADS consists of a total of 14 self-report items, divided into two subscales: seven related to anxiety and seven related to depression. Items are rated on a four-point Likert scale ranging from 0 to 3. Higher scores indicate more severe symptoms.
Sit-up Test | Baseline, at 8 week, at 12 week
  The "Sit-up Test" will be used to assess trunk endurance among participants. This test measures the strength and endurance of abdominal muscles. Participants will begin in a supine position with knees flexed at approximately 140 degrees, feet flat on the floor, legs slightly abducted, arms parallel to the trunk with palms facing downward. They will be instructed to perform sit-up movements by extending their arms forward and then returning to the starting position. The number of sit-ups completed within one minute will be recorded. Time will be tracked using a stopwatch. The validity and reliability of remote application of this test have been established.
Modified Push-up Test | Baseline, at 8 week, at 12 week
  The "Modified Push-up Test" will be conducted to assess trunk endurance. Participants will assume a prone position with hands positioned at shoulder level, elbows flexed, and the body aligned to allow for elbow extension and flexion. They will be asked to lift their head, shoulders, and trunk off the ground by fully extending their elbows and to repeat this movement for 40 seconds. The number of completed push-ups within this duration will be recorded. The validity and reliability of remote application of this test have been confirme.
Plank Test | Baseline, at 8 week, at 12 week
  The "Plank Test" will be used to evaluate trunk endurance. Participants will be positioned in a prone posture, resting on their forearms and toes, with their pelvis elevated and their body forming a straight line parallel to the ground. They will be instructed to maintain this position for as long as possible. The duration (in seconds) until the participant can no longer hold the position will be recorded. The validity and reliability of remote application of this test have been verified.
Side Bridge Test | Baseline, at 8 week, at 12 week
  The "Side Bridge Test" will be used to assess trunk endurance. Participants will be instructed to lie on their side with their legs extended and the upper arm placed across the chest, touching the opposite shoulder. The supporting elbow will be flexed, allowing weight to be distributed through the elbow and forearm. Participants will be asked to lift their hips off the ground while maintaining a straight body alignment, supported by the elbow and feet. The test will end when the participant loses the correct posture, and the duration (in seconds) of holding the position will be recorded. This test will be performed bilaterally. The validity and reliability of remote application of this test have been confirmed.
Timed Up and Go Test | Baseline, at 8 week, at 12 week
  The "Timed Up and Go Test" will be used to assess participants' functional capacity. Participants will be asked to stand up from a chair with armrests, walk three meters, turn around, return to the chair, and sit down. The total time taken to complete this task will be measured. The validity and reliability of remote application of this test have been established.
30-Second Chair Stand Test | Baseline, at 8 week, at 12 week
  The "30-Second Chair Stand Test" will be used to assess participants' functional capacity. Participants will use a chair with a seat height of 45-47 cm, ensuring their feet are in contact with the ground. Beginning in a seated position with arms crossed over the chest, they will be asked to stand up and sit down as many times as possible within 30 seconds. The number of completed repetitions will constitute the test score. The participant must fully extend their hips and knees while standing. The validity and reliability of remote application of this test have been confirmed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No